CLINICAL TRIAL: NCT04737473
Title: General Anesthesia Usiing Fentanyl Plus Propofol Plus Rococuronium Plus Isoflurane Versus Ketamime Plus Magnesium Sulphate Plus Lidocaine Plus Clonidine Plus Propofol Plus Rococuronium Plus Isoflurane in Gynaecology Surgery
Brief Title: The Comparative Efficacy and Safety of Two General Anesthesia Protocols Consisting of Fentanyl Plus Propofol Plus Rococuronium Plus Isoflurane Versus Ketamime Plus Magnesium Sulphate Plus Lidocaine Plus Clonidine Plus Propofol Plus Rococuronium Plus Isoflurane for Gynaecology Surgery in Cameroon
Acronym: OFA-AFRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Joel Noutakdie Tochie, Medical Doctor/Anesthetist, University of Yaounde 1
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: UY1
Record Dates: First submitted 2021-01-03; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Opioids; Clinical Trial; Anesthesia; Gynecology; Surgery
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opiod Free Anesthesia (OFA) group (Experimental): The OFA protocol will entailed induction of anesthesia intravenously by the administration of the following drugs: magnesium sulfate 40mg/kg (without exceeding 2.5g), lidocaine 1.5mg/kg, ketamine 25mg, propofol 1.5-2mg/kg, dexamethasone 8mg and rocuronium 0.6mg/kg. Anesthesia will be maintained using isofluorane through volume controlled ventilation, and a mixture of magnesium sulfate 40mg/kg (without exceeding 2.5g/24h), lidocaine 1.5mg/kg, ketamine 25mg, and clonidine 1ug/kg in an electric pump syringe at 10 - 15 ml/h.
  Interventions: Drug: Opiod Free Anesthesia
- General anesthesia (GA) group (Active Comparator): The GA protocol described in the intervention arm
  Interventions: Drug: Opiod Free Anesthesia

INTERVENTIONS:
Drug: Opiod Free Anesthesia — The OFA protocol will entailed induction of anesthesia intravenously by the administration of the following drugs: magnesium sulfate 40mg/kg (without exceeding 2.5g), lidocaine 1.5mg/kg, ketamine 25mg, propofol 1.5-2mg/kg, dexamethasone 8mg and rocuronium
  Other Names: General anesthesia (GA)

SUMMARY:
Recently, a lot of side effects have been identified from the perioperative use of opioids. To remedy this, anesthesia research has recently focused on providing safe general anesthesia without opioids in a new concept or anesthetic technic called Opiod Free Anesthesia (OFA). Evidence on the effectiveness and safety of OFA is scarce in Africa, with no report from Cameroon.The aim of this study is to demonstrate the feasibility of an adapted OFA protocol as well as its efficacy and safety in very painful surgeries like gynaecology surgery in a low-resource setting.

DETAILED DESCRIPTION:
The investigators intend to conduct a single-blinded randomized controlled trial on American Society of Anesthesiologists (ASA) I and II women who will undergo elective myomectomy, hysterectomy, ovarian cystectomy and mastectomy between June 2021 to September 2021 at the Yaounde Gynaeco-Obstetric and Pediatric Hospital of Cameroon. Participants will be matched for age and parity in a ratio of 1:1 into an Opiod Free Anesthesia (OFA) group and a general anesthesia (GA) group. The primary endpoints shall be the success rate of OFA. The secondary endpoints shall be the mumber or frequency of postoperative complications like respiratory distress, nausea and vomiting, paralitic ileus and severe postoperative pain. The threshold for statistical significance will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria :

* American Society of Anesthesiology (ASA) grade I and II patients
* Patients undergoing an elective myomectomy, hysterectomy, ovarian cystectomy or total mastectomy.
* Patients who will be operated for benign pathologies or localized malignancies

Exclusion Criteria :

* Past history of allergy to any of the anesthetic drugs
* Refusal to consent to participate in the study

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females aged between 21 to 70 years old
Enrollment: 36 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-09-28 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
Intraoperative variables | 9 months
  The success rate of OFA (defined as no intraoperative administration of opioids).

SECONDARY OUTCOMES:
Postoperative variables | 9 months
  The number of postoperative complications in the OFA and GA group. The complications to be determined will be the bumber of occurrence of severe postoperative pain, nausea and vomiting, respiratory distress and paralytic ileus

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Ze Minkande, MD, Study Director — University of Yaounde I
Locations (1):
- Yaounde Gynaeco-Obstetric and Pediatric Hospital, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guinot PG, Spitz A, Berthoud V, Ellouze O, Missaoui A, Constandache T, Grosjean S, Radhouani M, Anciaux JB, Parthiot JP, Merle JP, Nowobilski N, Nguyen M, Bouhemad B. Effect of opioid-free anaesthesia on post-operative period in cardiac surgery: a retrospective matched case-control study. BMC Anesthesiol. 2019 Jul 31;19(1):136. doi: 10.1186/s12871-019-0802-y. PMID 31366330
- [Result] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933
- [Derived] Tochie JN, Bengono Bengono RS, Metogo JM, Ndikontar R, Ngouatna S, Ntock FN, Minkande JZ. The efficacy and safety of an adapted opioid-free anesthesia regimen versus conventional general anesthesia in gynecological surgery for low-resource settings: a randomized pilot study. BMC Anesthesiol. 2022 Oct 24;22(1):325. doi: 10.1186/s12871-022-01856-6. PMID 36280804